CLINICAL TRIAL: NCT00996866
Title: Vitamin D Supplementation Requirement in Obese Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enable to further recruit study subjects
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08028
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Half of subjects will be randomized to the placebo group.
  Interventions: Drug: placebo
- Vitamin D3 (Active Comparator): This is the study group that receives Vitamin D supplementation.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D supplementation will follow an algorithm for initial vitamin D dosing and for dose changes. Subjects will receive 100 ug/day of vitamin D3 if their 25(OH)D level is less than 50nmol/L and 50 ug/day if their 25(OH)D level is between 50 and 80 ug/day.
  Arms: Vitamin D3
Drug: placebo — The placebo group will receive sugar pills appearing similar to the vitamin D capsules.
  Arms: Placebo

SUMMARY:
Vitamin D deficiency is common in obese patients. Most of vitamin D supplementation studies were done with non-obese subjects. This study looks at vitamin D supplementation requirements in obese patients as compared to non-obese subjects. This study also looks at changes in vitamin D level in obese patients undergoing medical weight loss. It is thought that obese patients have vitamin D deficiency through storage of vitamin D in the fat compartment not readily available for blood measurement. The investigators' hypothesis is that with medical weight loss vitamin D levels will increase in obese subjects.

DETAILED DESCRIPTION:
We intend to study changes in serum 25(OH)D level with calorie restricted weight loss in obese subjects. This will be a double dummy, placebo controlled randomized trial. Subjects whose serum 25(OH)D level is below 80 nmol/L will be assigned randomly to either the vitamin D supplemented or the placebo group. Those who are assigned to the placebo group will be weighed on a weekly basis and serum 25(OH)D level will be followed every 8 weeks for a minimum of 16 weeks and extended to the duration of weight loss along with serum calcium level. Changes in serum 25(OH)D level will be obtained with weight loss through restricted caloric intake.

To study the 25(OH)D dose-response curve with vitamin D supplementation in obese subjects, vitamin D supplemented group will receive initial daily vitamin D3 supplementation dose based on their baseline serum 25(OH)D level as described in Methods and Procedures section. Serum 25(OH)D levels will be drawn at 8 weeks and adjustments to the dose will be made based on the an algorithm to achieve serum 25(OH)D levels between 80 and 140 nmol/L. The dose-response curve obtained at 8 weeks will be compared to the one already established with non-obese subjects. Serum 25(OH)D level will be obtained at 16 weeks and compared with the data available from non-obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between the ages of 18 and 70 years old who are enrolled in our Weight Management Program with baseline BMI > 30 Kg/m2.

Exclusion Criteria:

* Pregnancy,
* Serum 25(OH)D level greater than 80 nmol/L,
* Hypercalcemia (serum calcium level greater than the upper limit of normal),
* Recent surgery or illness,
* Those with chronic use of medications that influence calcium/vitamin D metabolism such as anti-convulsants, lithium and steroids. Thiazide diuretics for hypertension will be acceptable.
* Subjects with sarcoidosis will be excluded.
* Those who do not qualify to participate in the Weight Management Program will be excluded. They include subjects with active substance abuse and unstable cardiac disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Aloia,, MD, Principal Investigator — Winthrop-Unviersity Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited during the winter months from areas in a surrounding Long Island, New York by advertisement through flyers and direct mail. Volunteers were 18-65 years old with a BMI of >35kg/m2. Recruitment began in January of 2009 at the Bone Mineral Research Center at Winthrop University Hospital
Pre-assignment Details: Participants underwent a comprehensive history and physical examination and provides a blood specimen for laboratory measurements at baseline. Participants with 25(OH)D greater or equal to 80nmol/L at baseline were excluded from the study. The anticipated enrollment of 39 was an error.
Period: Overall Study
Arm/Group | Placebo | Vitamin D3
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D3 | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (7.43) | 53.5 (12.5) | 54.8 (9.83)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 5 | 8 | 13
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Level of 25(OH)D
Description: Vitamin D (25(OH)D) level at Baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 13 | 11
nmol/L | 51.1 (13.9) | 49.2 (15.3)

2. Primary Outcome: Mean Level of 25(OH)D
Description: Vitamin D (25(OH)D) level at Month 2.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 13 | 11
nmol/L | 49.9 (17.9) | 74.5 (13.43)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date the patient started the study medications until the date they completed the study, typically 2 months.
Arm/Group | Placebo | Vitamin D3
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes